CLINICAL TRIAL: NCT02655549
Title: A Phase 1a Double-Blind, Randomized, Placebo-Controlled, Dose-Escalation Study Assessing Safety and Immunogenicity of Px563L and RPA563 Administered by Intramuscular Injection in Healthy Adult Volunteers
Brief Title: A Study of Anthrax Vaccines Px563L and RPA563 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfenex, Inc (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PF563-101
Record Dates: First submitted 2016-01-12; First posted 2016-01-14 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Anthrax
MeSH Terms: conditions — Anthrax

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 of Px563L, RPA563, or placebo (Experimental): Intramuscular injections of Px563L, RPA563, or placebo
  Interventions: Biological: Px563L, RPA563, or placebo
- Cohort 2 of Px563L, RPA563, or placebo (Experimental): Intramuscular injections of Px563L, RPA563, or placebo
  Interventions: Biological: Px563L, RPA563, or placebo
- Cohort 3 of Px563L, RPA563, or placebo (Experimental): Intramuscular injections of Px563L, RPA563, or placebo
  Interventions: Biological: Px563L, RPA563, or placebo

INTERVENTIONS:
Biological: Px563L, RPA563, or placebo — Two intramuscular injections

SUMMARY:
The trial investigates Px563L and RPA563, two formulations of a novel anthrax vaccine.

DETAILED DESCRIPTION:
This is a Phase 1, double-blind, randomized, placebo-controlled study to evaluate the safety, tolerability, and immunogenicity of Px563L or RPA563 administered intramuscularly. All subjects will be followed for safety and tolerability for 393 days after the initial vaccination. Immunogenicity analyses will be performed for up to 182 days, including an interim analysis based on Day 70 results, after the initial vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to read and understand the consent process and sign an informed consent form (ICF).
* Females or males between the ages of 18 and 55, inclusive, at the time of informed consent.
* Healthy or with stable medical conditions not requiring continuous medication.

Exclusion Criteria:

* Female subjects who are pregnant or breastfeeding.
* A history of anthrax disease or receipt of an anthrax vaccine at any time in the past, exposure to or infection with B. anthracis, or has received any investigational anthrax vaccine or treatment (e.g., monoclonal antibodies, anthrax immune globulin).
* Positive test for human immunodeficiency virus (HIV), hepatitis C or hepatitis B (surface antigen).
* History of any malignant neoplasm or receipt of anti-neoplastic agents within the last 5 years, with the exception of adequately treated, localized or in situ non-melanoma of the skin (e.g., basal cell carcinoma) or of the cervix.
* History of immunodeficiency, chronic illness requiring continuous or frequent medical intervention, autoimmune disease, bleeding disorder, hemoglobinopathy, prior solid organ or bone marrow transplant, or any known history in the past 5 years of cardiac disease.
* Evidence of alcohol abuse (i.e., requiring treatment) or substance abuse (i.e., any use of illicit drugs) within 6 months prior to screening.
* History of severe allergy (e.g., anaphylaxis) to latex or rubber.
* Subjects who have significant scarring, tattoos, abrasions, rash, or other skin abnormality at the planned vaccination site that could interfere with evaluation of injection site..
* Use of any systemic steroids or other immunosuppressive agents within 2 years prior to screening; or use of topical, intranasal, or inhaled corticosteroids for ≥10 consecutive days within 1 year prior to screening.
* Administration of any licensed vaccines within 30 days prior to screening.
* History of anaphylaxis or other serious adverse reaction to vaccines.
* Donation or loss of >500 mL of blood or donation of plasma within 2 months of screening, or recipient of blood or blood products within 2 months of screening.
* Present or former member of US military or reservist who may have or will receive the licensed anthrax vaccine, or who has served in any military arena from January 1990 through present time.
* May be at risk for exposure to anthrax or may be required to receive the licensed anthrax vaccine (e.g., postal workers).
* Has previously participated in any anthrax vaccine or anti-protective antigen (PA) monoclonal antibody clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Adverse events (AE) and adverse events of special interest (AESI) for vaccines | 393 days

SECONDARY OUTCOMES:
Anthrax toxin neutralizing antibody (TNA) 50% neutralization factor (NF50) value | 182 days

CONTACTS AND LOCATIONS:
Overall Officials: Barbara K Lomeli, M.D., Principal Investigator — Quintiles Phase One Services, LLC; Hubert C Chen, M.D., Study Director — Pfenex, Inc
Locations (1):
- Quintiles Phase One Services, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Schneider JC, Chen HC, Bautista E, Retallack D. Safety and immunogenicity of Px563L, a recombinant anthrax vaccine candidate, in a two-dose regimen for post-exposure prophylaxis in healthy adults. Vaccine. 2021 Oct 8;39(42):6333-6339. doi: 10.1016/j.vaccine.2021.08.075. Epub 2021 Sep 17. PMID 34544599